CLINICAL TRIAL: NCT01348568
Title: Effect of Low Glycemic Index Diets (With Canola Oil) on Glucose Control in Non-Insulin Dependent Diabetics
Brief Title: Low Glycemic Index Diet (With Canola Oil) for Type 2 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canola Council of Canada (Other)
Responsible Party: Principal Investigator, David Jenkins, Principle Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-191
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low glycemic index diet with canola oil bread (Experimental): Subjects will be given whole wheat bread which includes canola oil, and advised to follow a diabetic diet using low glycemic index foods.
  Interventions: Dietary Supplement: low glycemic index diet with canola oil bread
- high fiber diet (Active Comparator): Subjects will be given whole wheat bread, and advised to follow a healthy high fiber diabetic diet.
  Interventions: Dietary Supplement: High fiber diet

INTERVENTIONS:
Dietary Supplement: low glycemic index diet with canola oil bread
  Arms: Low glycemic index diet with canola oil bread
Dietary Supplement: High fiber diet
  Arms: high fiber diet

SUMMARY:
Healthy individuals with type 2 diabetes will receive intensive counseling on food selection to improve glucose control using either high cereal fiber dietary strategies or low glycemic index foods especially canola oil containing bread. The treatments will last 3 months with bloods taken for HbA1c, glucose and blood lipids. If the study shows a benefit for either or both diets, then use of high fiber, and/or low glycemic index foods with canola oil, may provide another potential way to improve glucose control and lower cholesterol levels in non-insulin dependent diabetes.

DETAILED DESCRIPTION:
Overall design

* Sample size justification: The sample size requirement was determined based on the ability to detect a HbA1c reduction of at least 0.4 units, significance of the test (α) of 0.05, β of 2 and power (1-β) of 0.80 (The FDA criterion for drug effectiveness is a HbA1c reduction of 0.3 to 0.4 units). Examination of recent study results for HbA1c of the research group on type 2 diabetic subjects indicated a standard deviation of 0.32. So the desired total number to complete this study is N=80, or 120 enrolled assuming a 30% attrition rate.
* Design: All subjects will be randomized to one of two 12-week treatments in a two-treatment parallel design. Treatments: 1) low glycemic index dietary advice (e.g. to eat intact grain cereals, Pita Break Finland Rye and Little Stream Quinoa breads, parboiled rice, cracked wheat, pasta, peas, beans, lentils, and baked goods made from legume flour), with particular emphasis on a canola oil containing bread; and a 2) high cereal fiber diet emphasizing whole grains.

Duration: The study will consist of approximately two months recruitment and patient selection, and a 3 month treatment period.

Study Details: Fasting blood samples are obtained at screening, week -2, 0, 2, 4, 8, 10 and 12 of each study period for glucose, lipids and oxidation products. HbA1c will be assessed on all visits except week 2. Twenty-four hour urine for urinary C-peptide, isoprostane, urea, creatinine and electrolyte analyses will be obtained immediately prior to the beginning of the study and at the end of the 12 week treatment. At weeks 0 (baseline) and 12, endothelial function will be assessed. Following the 12 week treatment period, subjects who wish to undertake the alternate treatment will be given appropriate instruction.

* Setting: Risk Factor Modification Center at St. Michael's Hospital.
* Participants/controls (selection and inclusion/exclusion criteria):

Patient Selection: Healthy non-insulin dependent diabetic men and women will be recruited by newspaper advertisement, physician referral and the diabetic clinic at St. Michael's Hospital.

* Interventions: Diets: Diets will be the subjects' diabetic diets modified as above. Diet histories will be recorded at weeks 0, 2, 4, 8, 10 and 12. These diets will be assessed for consistency by the dietitian in the subject's presence. Where necessary, modifications in diet will be made to ensure weight maintenance.
* Privacy protection Subjects will have their data de-identified. Any databases with personal health information will be password protected. Also, patient data that has personal health information (e.g. patient charts) will be kept in locked cabinets, with the door locked to the room with the cabinets, and the centre door locked after 6 pm.
* Confidentiality of data All subjects will be assigned an identification code to ensure confidentiality. All data entered into files will use the identification codes. Access to data files will be limited to the PI, statisticians, dietitians, students, and data entry personnel working on the project.

The data obtained from the Endo-PAT test will be sent to a private statistical consultant in the United States for analysis. The dataset will be de-identified and only the statistical consultant and the research team will have access to this dataset.

-Identifiable data Subjects will be primarily identified by a code (number and letter) assigned by the study statistician. A separate chart with routine clinical information is maintained for contact with participants' family physicians.

DATA ANALYSIS:

a. Analysis method, including types of statistical or qualitative methods Results will be expressed as means ± standard error. The differences between treatment means will be assessed using the CONTRAST statement in SAS (Statistical Analysis Software) using -2 and zero bloods as baseline to calculate change and weeks 8, 10 and 12 for the CONTRAST. Pearson's correlations will be used to assess relationships between dietary compliance and weight reductions with blood lipid changes.

For Optional Sub-study:

In our recent diabetes study which looked at the effect of mixed nuts on blood sugar control (REB# 06-274), 44.8 % (35/78) of participants continued onto follow-up and 24% (19/78) completed follow-up. All crossed from either the muffin (control) or half dose nut supplement to the full dose nut (test) supplement. In a recent Portfolio study (REB#04-056), after 24 weeks 62.5% of participants crossed from DASH diet (control) to Portfolio diet (test). Assuming that in this study participants will also cross from the control diet to the test diet, we will use a paired t-test with no adjustment for baseline or sequence, as this is not a true crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with type 2 diabetes who

  * are treated with oral hypoglycemic agents at a stable dose for at least 8 weeks
  * have a HbA1c in the range of 6.5 to 8.5% at the initial screening visit and at the prestudy visit (visit just prior to randomization)
  * have diabetes diagnosed >6 months
  * have maintained stable weight for 2 months (within 3%)
  * have a valid OHIP card and a family physician
  * if prescribed lipid medication, have taken a stable dose for at least 2 weeks
  * if prescribed blood pressure medication, have taken a stable dose for at least 1 week
  * can keep written food records, with the use of a digital scale

Exclusion Criteria: Individuals who

* take insulin
* take steroids
* have GI disease (gastroparesis, celiac disease, ulcerative colitis, Crohn's Disease, IBS)
* have had a major cardiovascular event (stroke or myocardial infarction) in the past 6 months
* take warfarin (Coumadin)
* have had major surgery in the past 6 months
* have a major debilitating disorder
* have clinically significant liver disease (AST or ALT > 130 U/L), excluding NAFL or NASH
* have hepatitis B or C
* have renal failure (high creatinine > 150 mmol/L)
* have serum triglycerides ≥ 6.0 mmol/L
* have a history of cancer, except non-melanoma skin cancer (basal cell, squamous cell)
* have food allergies to canola oil, study food components
* have elevated blood pressure (> 145/90) unless approved by General Practitioner (GP)
* have acute or chronic infections (bacterial or viral)
* have chronic inflammatory diseases (e.g. rheumatoid arthritis, lupus; ulcerative colitis)
* have other conditions which in the opinion of any of the investigators would make them unsuitable for the study
* If HbA1c rises above 8.5% over two consecutive routine measurements, subjects will be referred back to their family doctors for an increase in anti hyperglycemic medications according to a predetermined protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
change in serum lipids | from prestudy and week 0, to end of treatment weeks 8, 10, and 12

SECONDARY OUTCOMES:
fasting glucose | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
change in weight, waist, and hip circumference | weeks 0 to 12
change in blood pressure | from prestudy and week 0, to end of treatment weeks 8, 10, and 12
creatinine, urea, and c-peptides in 24 hour urine collection | 0, 12 weeks
endothelial function | week 0, 12
cancer cell proliferation (in vitro) | week 0, 12

CONTACTS AND LOCATIONS:
Overall Officials: David J A Jenkins, MD, DSc, Principal Investigator — Dept of Nutritional Science, University of Toronto, Toronto, ON, Canada; Cyril W C Kendall, PhD, Principal Investigator — Dept of Nutritional Science, University of Toronto, Toronto, Canada; Robert Josse, MD, Principal Investigator — Dept of Medicine, Div of Endocrinology and Metabolism, St. Michael's, Toronto, ON, Canada
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins DJ, Kendall CW, Vuksan V, Faulkner D, Augustin LS, Mitchell S, Ireland C, Srichaikul K, Mirrahimi A, Chiavaroli L, Blanco Mejia S, Nishi S, Sahye-Pudaruth S, Patel D, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Josse RG, Leiter LA. Effect of lowering the glycemic load with canola oil on glycemic control and cardiovascular risk factors: a randomized controlled trial. Diabetes Care. 2014 Jul;37(7):1806-14. doi: 10.2337/dc13-2990. Epub 2014 Jun 14. PMID 24929428